CLINICAL TRIAL: NCT01263028
Title: Effects of Ergocalciferol on Erythropoetin Stimulating Agent Dose
Acronym: EASY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Strong enrollment efforts resulted in few eligible subjects and high screen failures due to CKD patients with higher vitamin D levels than anticipated.
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM2010001
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2012-09-20 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease Stages 3-5

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ergocalciferol supplementation (Experimental)
  Interventions: Drug: Ergocalciferol supplementation

INTERVENTIONS:
Drug: Ergocalciferol supplementation — Vitamin D in the form of ergocalciferol will be the drug utilized in the study. This medication is a Vitamin D analog and is normally used in the current study population to help augment those who are deficient in Vitamin D.

SUMMARY:
Hypothesis: The supplementation of Ergocalciferol (Vitamin D2) to those with Vitamin D deficiency in the Chronic Kidney Disease population requiring recombinant human erythropoietin for the treatment of anemia related to kidney disease will reduce the dose of erythropoietin required to maintain a nonanemic state.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease
* Age: >18yo
* Stable Hemoglobin (Hgb) for 1 month on stable dose of erythropoietin for 1 month (defined as erythropoietin dose within 15% of previous months erythropoietin dose)
* Unchanged maintenance oral or intravenous (IV) iron therapy for 1 month
* Serum 25-hydroxy Vitamin D levels < 30 ng/mL
* History of 25-hydroxy Vitamin D levels < 30 ng/mL currently on ergocalciferol replacement

Exclusion Criteria:

* On hemodialysis
* Chronic kidney disease 5
* Hypercalcemic (Calcium level > 11mg/dL)
* Pregnant female
* Iron deficient (iron saturation < 20%, Ferritin < 100ng/mL)
* Presence of active malignancy
* Presence of active infections
* Presence of active inflammatory properties
* Presence of blood dyscrasias
* Active bleeding or bleeding within the past 3 months (other than menses)
* B12 deficiency
* Folate deficiency
* Blood transfusion during participation
* Parathyroid levels exceeding the expected levels allowed for the stage of a subjects Chronic kidney disease (Target Parathyroid in: Chronic kidney disease 3 35-70 pg/mL, Chronic kidney disease 4 70-110 pg/mL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Sim, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Los Angeles Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in February 2011 at Kaiser Permanente Los Angeles Medical Center. Despite strong enrollment efforts only 6 particiants were enrolled out of 10 screened.
Pre-assignment Details: Participants were assessed for study inclusion based on chronic kidney disease (CKD) stage, age, current vitamin D levels <30 ng/ml as well as history of vitamin D levels < 30, and stable dose of erythropoietin and iron.
Period: Overall Study
Arm/Group | Ergocalciferol Supplementation
Started | 6
Completed | 0
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Study terminated due to low enrollment. | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ergocalciferol Supplementation
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Evaluate if Ergocalciferol Supplementation to Achieve 25-hydroxy Vitamin D Levels > 40ng/ml Will Decrease Erythropoietin Requirements
Time Frame: 24 Weeks
Groups:
- Ergocalciferol Supplementation: Ergocalciferol will be administered as 50,000 international units (IU) weekly regardless of Serum 25-hydroxy Vitamin D levels for 12 weeks. Then 50,000 IU every other week. If 25-hydroxy Vitamin D levels are below goal of 40ng/ml, subjects will continue on 50,000 IU ergocalciferol weekly until levels of 40ng/ml, are achieved.
Arm/Group | Ergocalciferol Supplementation
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Inflammatory Markers
Time Frame: 24 Weeks
Arm/Group | Ergocalciferol Supplementation
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Calcium, Phosphorous,Calcium x Phosphorous Product, and Parathyroid Hormone Levels
Time Frame: 24 Weeks
Arm/Group | Ergocalciferol Supplementation
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Iron Supplementation
Time Frame: 24 Weeks
Arm/Group | Ergocalciferol Supplementation
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Erythropoietin Adjusted for Change in Inflammatory Markers, Vitamin D Levels and Clinical and Demographic Confounders
Time Frame: 24 Weeks
Arm/Group | Ergocalciferol Supplementation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 36 Weeks
Arm/Group | Ergocalciferol Supplementation
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergocalciferol Supplementation (N=6)
Low Hemoglobin (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated due to insufficient enrollment numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes